CLINICAL TRIAL: NCT00278460
Title: A Phase II Study of Taxotere and Gemcitabine for Stages III-B and IV Non-Small Cell Lung Cancer
Brief Title: Gemcitabine and Docetaxel in Treating Patients With Recurrent Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000462116; CCCWFU-62199; AVENTIS-CCCWFU-62199; AG-CCCWFU-62199; CCCWFU-BG99-322
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer; recurrent non-small cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: docetaxel — 40 milligrams per meter squared infused over 30 minutes on day 1 and 8, repeated every 21 days
Drug: gemcitabine hydrochloride — 800 milligrams per meter squared intraveneously for two consecutive weeks followe by one week of no treatment then repeated.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with docetaxel works in treating patients with recurrent stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate of patients with recurrent stage IIIB and IV non-small cell lung cancer treated with gemcitabine hydrochloride and docetaxel.
* Determine the overall and progression-free survival of patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.

Secondary

* Determine the duration of response in patients treated with this regimen.

OUTLINE: Patients receive gemcitabine hydrochloride IV over 30 minutes followed by docetaxel IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for survival.

PROJECTED ACCRUAL: A total of 51 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IIIB or IV non-small cell lung cancer, including any of the following types:

  * Squamous cell carcinoma
  * Adenocarcinoma, including bronchoalveolar cell adenocarcinoma
  * Large cell anaplastic carcinoma, including giant and clear cell carcinomas
* Histologic or cytologic documentation of recurrence is required
* Measurable or evaluable disease, defined as any mass reproducibly measurable in 2 perpendicular diameters by physical examination or imaging

  * The following lesions are not considered measurable or evaluable:

    * Bone disease only
    * Pleural or pericardial effusions
    * Previously irradiated lesions, unless subsequent progression is documented
* CNS metastases allowed provided the patient undergoes at least 2 weeks of radiotherapy prior to study entry

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Negative pregnancy test
* CALGB performance status ≤ 1
* Life expectancy ≥ 3 months
* Granulocyte count > 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 2 times normal
* Bilirubin normal
* SGOT and/or SGPT ≤ 2.5 times upper limit of normal (ULN) AND alkaline phosphatase ≤ 1.5 times ULN OR
* Alkaline phosphatase 4 times ULN and SGOT and/or SGPT normal
* Ejection fraction normal by ECHO or MUGA
* No history of congestive heart failure
* No psychiatric illness that would preclude study compliance
* No serious medical or psychiatric illness that would preclude giving informed consent or limit survival to < 3 months
* No active uncontrolled bacterial, fungal, or viral infection
* No other malignancy within the past 5 years except curatively treated carcinoma in situ of the cervix or breast, basal cell or squamous carcinoma of the skin, or other surgically resected non-recurrent primary tumor not treated with adjuvant radiotherapy or chemotherapy
* No pre-existing peripheral neuropathy ≥ grade 2

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior major surgery and recovered from acute effects
* At least 2 weeks since prior palliative radiotherapy and recovered from acute toxic effects

  * Any persistent toxicity (e.g., alopecia or hyperpigmentation) not associated with clinical morbidity allowed
* No prior chemotherapy
* No concurrent cranial or thoracic radiation therapy
* No concurrent cytotoxic or hormonal therapy
* Concurrent palliative radiotherapy allowed for relief of localized pain and obstruction

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2000-11; Primary Completion 2006-02 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
patient response rate to weekly taxotere and gemcitabine | 6 weeks

SECONDARY OUTCOMES:
Evaluate toxicity of weekly Taxotere and Gemcitabine | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonius A. Miller, MD, Study Chair — Wake Forest University Health Sciences